CLINICAL TRIAL: NCT00654849
Title: Electrosurgical Bipolar Plasmakinetic Vessel Sealing During Abdominal Hysterectomy: A Randomized Controlled Trial
Acronym: PKAHRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Concentracion Norte de Petroleos (Other Government)
Responsible Party: Carlos Humberto Briones Landa MD, Servicios de Salud Petroleos Mexicanos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKHTA2007; PKHTA12345
Record Dates: First submitted 2008-04-02; First posted 2008-04-09 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Abdominal Hysterectomy for Benign Disease
Keywords: Electrosurgery; Gyrus Pk; abdominal hysterectomy; Blood Loss, Surgical; Length of stay; Overall cost
MeSH Terms: conditions — Hyperthermia; Blood Loss, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): compare security and effectiveness of use Electrosurgical Bipolar Plasmakinetic Vessel Sealing
  Interventions: Procedure: Plasmakinetic bipolar energy forceps
- 2 (Active Comparator): traditional abdominal hysterectomy technique with the use of sutures
  Interventions: Procedure: Abdominal Hysterectomy with traditional suture technique

INTERVENTIONS:
Procedure: Plasmakinetic bipolar energy forceps — Use of bipolar plasmakinetic vessel sealing during abdominal hysterectomy
  Other Names: Gyrus PK 3103PK
  Arms: 1
Procedure: Abdominal Hysterectomy with traditional suture technique — The abdominal hysterectomy was realized using sutures in the haemostasia of pedicles.
  Other Names: Traditional technique
  Arms: 2

SUMMARY:
Objective: To compare the safety and efficacy of the use of bipolar plasmakinetic vessel sealing (Gyrus Pk) usage versus standard technique when performing total abdominal hysterectomy for benign disease.

Material and Methods: controlled randomized trial involving 94 women who underwent total abdominal hysterectomy. 47 procedures were performed using bipolar plasmakinetic vessel sealing and the remaining 47 with the standard sutures technique. The primary outcomes were improvement in terms of blood loss, procedure time, length of hospital stay, and overall cost of the procedure. Statistical methodology considered significant P <0.05.

DETAILED DESCRIPTION:
All patients were right-holders of the Petroleos Mexicanos (Mexican oil company) medical network who required hysterectomy surgical treatment for benign causes All patients included in the study signed an informed consent form, knowing all possible implications of the procedure Patients were randomly assigned to one of the two techniques: 1. plasmakinetic bipolar energy forceps (Gyrus PK) and 2. Standard technique using sutures The surgical steps other than placement of suture are identical to those used during standard abdominal hysterectomy. Time of the procedure was considered from the moment skin was first cut-open, until it was fully closed, previously checking satisfactory homeostasis.

Blood loss was estimated by the anesthesiology service. Further data compiled included time spent in hospital and the total cost of the procedure.

Post-surgery complications were recorded at the follow up visits one and 4 weeks after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a benign disease as indication for hysterectomy

Exclusion Criteria:

* Hysterectomy for malignant pathology
* Laparoscopic or vaginal hysterectomy
* Any patient in which the procedure used both techniques
* Obstetric hysterectomy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Blood loss measured by anesthesiology service during the procedure | 1 year

SECONDARY OUTCOMES:
Operating time | 1 year
Length of stay | 1 year
The total cost of the procedure | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Carlos H Briones, MD, Principal Investigator — Servicios Medicos de Petroleos Mexicanos
Locations (1):
- Hospital Central Norte, Distrito Federal, Mexico

REFERENCES:
- [Background] Farquhar CM, Steiner CA. Hysterectomy rates in the United States 1990-1997. Obstet Gynecol. 2002 Feb;99(2):229-34. doi: 10.1016/s0029-7844(01)01723-9. PMID 11814502
- [Background] Broder MS, Kanouse DE, Mittman BS, Bernstein SJ. The appropriateness of recommendations for hysterectomy. Obstet Gynecol. 2000 Feb;95(2):199-205. doi: 10.1016/s0029-7844(99)00519-0. PMID 10674580
- [Background] Presthus JB, Brooks PG, Kirchhof N. Vessel sealing using a pulsed bipolar system and open forceps. J Am Assoc Gynecol Laparosc. 2003 Nov;10(4):528-33. doi: 10.1016/s1074-3804(05)60161-2. PMID 14738643
- [Background] Hagen B, Eriksson N, Sundset M. Randomised controlled trial of LigaSure versus conventional suture ligature for abdominal hysterectomy. BJOG. 2005 Jul;112(7):968-70. doi: 10.1111/j.1471-0528.2005.00561.x. PMID 15958001
- [Background] Dessole S, Rubattu G, Capobianco G, Caredda S, Cherchi PL. Utility of bipolar electrocautery scissors for abdominal hysterectomy. Am J Obstet Gynecol. 2000 Aug;183(2):396-9. doi: 10.1067/mob.2000.105911. PMID 10942476
- [Background] Rock J.,Howards WJ. Histerectomía em: Te Linde Ginecologia Quirúrgica .9ed,Editorial Panamericana Argentina 2006 (31):875-896. Uterine Surgery, En Nezhat C., Nezhat F., Luciano A., et al, eds., operative Gynecologic Laparoscopy; 1ª Ed: New York, New York; McGraw Hill, Inc.: 1995; 216-38. Hernández-Denis A. Audifred-Salomón J. Aspectos Generales en Endoscopia. En Hernández-Denis A. Audifred-Salomón J. Manual de Endoscopica en Ginecología. México; 2005:5-23.